CLINICAL TRIAL: NCT01024868
Title: Assessment of Spread of Transversus Abdominis Plane Block After Administration of 20 ml Ropivacaine 0,5% Bilaterally
Brief Title: Assessment of Spread of Transversus Abdominis Plane Block
Status: Completed | Type: Observational
Sponsor: Herlev Hospital (Other)
Collaborators: Glostrup University Hospital, Copenhagen (Other)
Responsible Party: Dr Anja U. Mitchell, Herlev University Hospital, Copenhagen
Other Study IDs: TDTSG-1
Record Dates: First submitted 2009-12-02; First posted 2009-12-03 (Estimated); Last update posted 2010-05-04 (Estimated); Status verified 2009-12

CONDITIONS: Transversus Abdominis Plane Block
Keywords: Transversus Abdominis Plane Block

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- TAP block: Patients before undergoing laparoscopic or other abdominal surgery
  Interventions: Drug: Ropivacaine 0,5%

INTERVENTIONS:
Drug: Ropivacaine 0,5% — Injection of ropivacaine 0,5% 20 ml bilaterally before surgery

SUMMARY:
For the purpose of assessing the spread of the local anaesthetic after injecting it between abdominal muscles on both sides, the investigators will test if the patient can feel a change in the perception of cold and warm, as well as being pricked with a blunt needle. The investigators will also take several blood samples, together with routine samples, to measure the concentration of the local anesthetic in the blood.

ELIGIBILITY:
Inclusion Criteria:

* undergo abdominal surgery, eligible for TAP block, over 18, BMI 20-40

Exclusion Criteria:

* does not speak danish, does not consent, does not fulfill inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients undergoing abdominal surgery
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2009-12; Primary Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ann M Møller, dr. med., Study Director — Herlev Hospital
Locations (1):
- Herlev University Hospital, Herlev, Denmark

REFERENCES:
- [Derived] Torup H, Mitchell AU, Breindahl T, Hansen EG, Rosenberg J, Moller AM. Potentially toxic concentrations in blood of total ropivacaine after bilateral transversus abdominis plane blocks; a pharmacokinetic study. Eur J Anaesthesiol. 2012 May;29(5):235-8. doi: 10.1097/EJA.0b013e328350b0d5. PMID 22450529
- [Derived] Mitchell AU, Torup H, Hansen EG, Petersen PL, Mathiesen O, Dahl JB, Rosenberg J, Moller AM. Effective dermatomal blockade after subcostal transversus abdominis plane block. Dan Med J. 2012 Mar;59(3):A4404. PMID 22381092